CLINICAL TRIAL: NCT06431646
Title: Evaluation of the Effectiveness of Web-Based Education on Premenstrual Syndrome (PMS) Symptoms and Quality of Life
Brief Title: Effectiveness of Web-Based Education on Premenstrual Syndrome and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sevgi Özkan, Dean of Health Sciences Faculty, Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 60116787-020/31827; 2020SABE021 (Other Grant/Funding Number: PamukkaleU Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2024-05-15; First posted 2024-05-28 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-05

CONDITIONS: Premenstrual Syndrome; Quality of Life
Keywords: Premenstrual Syndrome; Web-Based; Nurse-Led; Health Education; Quality of Life
MeSH Terms: conditions — Premenstrual Syndrome; Health Education | interventions — Spectrometry, Fluorescence

STUDY DESIGN:
Intervention Model Description: Randomized controlled study with a pretest-posttest design
Who Masked: Participant
Masking Description: Student
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Web-based education with weekly updates about PMS (definition, symptoms, treatment etc.) and management (especially, non-pharmacologic strategies) for 4 weeks
  Interventions: Behavioral: A web-based education intervention developed for university students with PMS
- Control Group (No Intervention): No special intervention

INTERVENTIONS:
Behavioral: A web-based education intervention developed for university students with PMS — The web-based education program includes the definition, prevalence, importance, causes, symptoms, diagnosis, risk factors, management strategies and treatment options of PMS. The education emphasizes non-pharmacological strategies for managing PMS, including diet, exercise and body mass index (BMI), sleep hygiene, smoking cessation, stress management, as well as vitamin and mineral supplements, herbal therapy, acupuncture, acupressure and reflexology.
  Other Names: Premenstrual Syndrome Education Program
  Arms: Intervention Group

SUMMARY:
Digital solutions are becoming increasingly prevalent, addressing health concerns through innovative means has become imperative. Among these concerns, Premenstrual Syndrome (PMS) stands out as a significant challenge that affecting the physical and emotional well-being of women of reproductive age. Despite previous studies demonstrating the effectiveness of health education for PMS, there remains a gap in providing accessible and evidence-based interventions. The present study aims to fill this gap leveraging technology to deliver targeted information and support to women. For this reason, the purpose of this randomized controlled trial is to evaluate the effectiveness of a web-based health education in university students with PMS. The main questions it aims to answer are:

* Does web-based education lower the premenstrual symptoms in university students with PMS?
* Does web-based education improve the quality of life in university students with PMS?

Researchers compared web-based education to a control (no special intervention) to see if intervention works to management PMS. Intervention group participants received web-based education with weekly updates about PMS (definition, symptoms, treatment etc.) and management strategies for 4 weeks.

DETAILED DESCRIPTION:
The study was planned as a parallel, single-blind, randomized, controlled experimental study with a pretest-posttest design. The sample group of the research was the nursing department of a Faculty of Health Sciences in Pamukkale University. Eligibility was determined by the Premenstrual Syndrome Scale and personal information form. The sample size was calculated in the PS Power and Sample Size Calculations 3.1.6 program by using data from a previous study with a large effect size (α =0.05, d=0.86). Accordingly, it was found that at least 32 participants should be taken for each group to sampling for 80% power. To avoid possible data loss, all participants (n=74) determined to be eligible were included in the study. A simple randomization method was used in this study. Outcomes were measured at baseline, 4 weeks, and 12 weeks after the intervention began. Data were collected using the Premenstrual Syndrome Scale, Premenstrual Symptoms Impact Scale, System Usability Scale, and personal information form.

ELIGIBILITY:
Inclusion Criteria:

* PMS (PMSS score of 132+)
* Normal menstrual cycle (21-35 days)
* No oral contraceptives
* No psychiatric problems or treatment
* Active Internet use
* Over 18
* Volunteering to participate in research

Exclusion Criteria:

* Internet access problems
* Website login issues
* Unanswered survey questions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female students with PMS
Enrollment: 67 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Premenstrual Syndrome Scale (PMSS) | Change from baseline score at 4 and 12 weeks
  The scale consists of 44 questions about experiences in the seven days before menstruation. Scores range from 44 to 220, with a total score above 132 indicating the presence of PMS. The scale contains nine subscales, each of which assesses a distinct aspect of PMS-related symptoms.
Premenstrual Symptoms Impact Scale (PMSIS) | Change from baseline score at 4 and 12 weeks
  The scale consists of six questions to evaluate the impact of PMS-related quality of life. Each question assesses the intensity of symptoms experienced during the "last premenstrual period". Total scores range from 6 to 30, with higher scores indicating worsening quality of life.

SECONDARY OUTCOMES:
System Usability Scale (SUS) | At the end of the 4-week intervention
  The scale consists of 10 questions to evaluate user satisfaction with system usability. The total score obtained from the scale is multiplied by 2.5, resulting in a score between 0 and 100. A score of 68 and above indicates that the system is usable.

OTHER OUTCOMES:
Personal Information Form | Baseline
  The form was designed by the researchers to collect students' socio-demographic characteristics and risk factors associated with PMS.

CONTACTS AND LOCATIONS:
Overall Officials: Ece Özkaradiğin, RN, MSc, Study Chair — Pamukkale University; Sevgi Özkan, RN, PhD, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Management of Premenstrual Syndrome: Green-top Guideline No. 48. BJOG. 2017 Feb;124(3):e73-e105. doi: 10.1111/1471-0528.14260. Epub 2016 Nov 30. No abstract available. PMID 27900828
- [Background] Taghizadeh Z, Shirmohammadi M, Feizi A, Arbabi M. The effect of cognitive behavioural psycho-education on premenstrual syndrome and related symptoms. J Psychiatr Ment Health Nurs. 2013 Oct;20(8):705-13. doi: 10.1111/j.1365-2850.2012.01965.x. Epub 2012 Sep 10. PMID 22957993
- [Background] Ayaz-Alkaya S, Yaman-Sozbir S, Terzi H. The effect of Health Belief Model-based health education programme on coping with premenstrual syndrome: a randomised controlled trial. Int J Nurs Pract. 2020 Apr;26(2):e12816. doi: 10.1111/ijn.12816. Epub 2020 Jan 27. PMID 31985138
- [Background] Simsek Kucukkelepce D, Timur Tashan S. The effects of health belief model-based education and acupressure for coping with premenstrual syndrome on premenstrual symptoms and quality of life: A randomized-controlled trial. Perspect Psychiatr Care. 2021 Jan;57(1):189-197. doi: 10.1111/ppc.12546. Epub 2020 May 29. PMID 32468669
- [Background] Borji-Navan S, Mohammad-Alizadeh-Charandabi S, Esmaeilpour K, Mirghafourvand M, Ahmadian-Khooinarood A. Internet-based cognitive-behavioral therapy for premenstrual syndrome: a randomized controlled trial. BMC Womens Health. 2022 Jan 8;22(1):5. doi: 10.1186/s12905-021-01589-7. PMID 34996424